CLINICAL TRIAL: NCT00968032
Title: Single-center Non-comparative, Prospective Interventional Clinical Investigation on the Procedural Success and Safety of the Nit-Occlud® PFO Closure Device and Its Application System.
Brief Title: Procedural Success and Safety of the Nit-Occlud® Patent Foramen Ovale (PFO) Closure Device and Its Application System
Acronym: 09k003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: pfm medical gmbh (Industry)
Collaborators: MDT Medical Device Testing GmbH (Industry)
Responsible Party: Christof Schmeer head of quality assurance pfm group, pfm medical ag
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09k003
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2011-03-09 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Foramen Ovale, Patent; Heart Catheterization; Heart Septal Defects, Atrial
Keywords: PFO; Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Nit-Occlud® PFO — Transcatheter implantation of a PFO occluder (Nitinol double Umbrella)

SUMMARY:
The foramen ovale is an opening in the interatrial septum. It results from an incomplete coverage of the ostium secundum. In 10 to 24% of the general population incomplete fibrosis of the interatrial septum is a clinical finding and is defined as a patent foramen ovale (PFO). The Nit-Occlud® PFO umbrella is a permanent implant for closing PFOs that is implanted in the PFO using minimally invasive catheter technology. The umbrella is made from Nitinol, a material with superelastic properties, which, in its relaxed state, has the form of a double umbrella. This is a single-center, non-comparative, prospective interventional clinical investigation involving 1 center in Germany to assess the effectiveness, safety and practicability of implantation of the Nit-Occlud PFO® Closure Device.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of patent foramen ovale (PFO)

1. Age between 18 and 65 years of both gender
2. Ability to give written informed consent after being told the potential benefits and risks of entering the trial to understand the planned clinical study and able to participate in all follow-up procedures
3. Signed informed consent
4. Presenting with neurological symptoms and at least one of the following clinical circumstances:

   * Diagnosis of cryptogenic stroke based on clinical neurological examination
   * Diagnosis of a transient ischemic attack (TIA) based on clinical neurological examination
5. PFO defect with or without atrial septal aneurysm of a balloon stretched diameter less than 18 mm. PFO tunnel length less than 10 mm in TEE
6. Mental and physical ability of patient to follow the protocol according to compliance to time schedule, treatment plan,completion of CRF pages and further study procedures.

Exclusion Criteria:

1. PFO dimensions exceeding Inclusion criterium 5)
2. Active endocarditis
3. Presence of an infectious disease
4. Vascular anatomy unable to accommodate the appropriate-sized sheath for device introduction
5. Current arrhythmia, or history of arrhythmia
6. Prior cardiac surgery, including implantation of active and non-active cardiac device (coronary stent is allowed)
7. Confinement to bed (because of higher potential for clot formation)
8. Heart abnormality other than PFO
9. Accessory atrial defects
10. Participation in an investigational drug or device trial within 30 days prior to selection, or current inclusion in any other clinical trial or research project
11. Known allergy to nickel
12. Known allergy to contrast agents
13. Cancerogenic disease or malignant tumor, or other severe disease
14. Intracardiac mass or vegetation
15. Thrombus at the intended site of implant or documented evidence of venous thrombus in the vessel to which access to the defect is gained
16. Unable to tolerate Aspirin or Clopidogrel, and/or antibiotic prophylaxis for at least three months following the procedure
17. Pregnant or breast feeding female patients
18. Subjects who, in the opinion of the investigator, will be inappropriate for inclusion into this trial or will not comply with requirements of the study
19. Subjects who are imprisoned (according to MPG § 20.3)
20. Patients who are lawfully kept in an institution

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, Prof. Dr., Principal Investigator — Cardio-Vascular Centre, Sankt Kathrinen, Frankfurt, Germany
Locations (1):
- Cardio-Vascular Centre, Sankt Kathrinen, Frankfurt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was set between June 2009 and July 2010 at a single medical clinic.
Pre-assignment Details: No enrolled participants were excluded from the trial.
Groups:
- Nit-Occlud® PFO Implantation Group: Patients suffering from PFO and suitable for closure of the defect with the Nit-Occlud® PFO Closure Device
Period: Overall Study
Arm/Group | Nit-Occlud® PFO Implantation Group
Started | 63
Completed | 61 (1 patient not receiving investigational device due to failure in usage 1 patient denied latest FU)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nit-Occlud® PFO
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 61
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 45.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 37
Region of Enrollment [Number; unit: participants]
  Germany | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Successful Implantation.
Description: The implantation of the device under investigation in a single patient is defined as successful if delivery, placement and release of the device in a stable position is successful. The value will be compared to the number of patient enrolled.
Time Frame: 6 weeks ± 2 weeks
Measure: Number; unit: participants
Arm/Group | Nit-Occlud® PFO
Number analyzed (Participants) | 63
participants | 62

ADVERSE EVENTS:
Time Frame: Adverse Events were observed for each patient during a 6 week FU period (6 weeks +- 2 weeks). Adverse events were judged by the relationship to the investigational device
Description: No AE led to discontinuation of the study. Causal relationship to the device was not ruled out in 19 AEs. Within these, for 15 AEs the relationship was recorded as unknown, 2 AEs were recorded as possibly related, and 2 AEs were recorded as related. All device related AEs were reported as of mild intensity.
Arm/Group | Nit-Occlud® PFO
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 19/63
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nit-Occlud® PFO (N=63)
Cardiac General (Cardiac disorders) | 5 (5)
Neurology (Nervous system disorders) | 4 (4)
Cardiac Arrhythmia (Cardiac disorders) | 3 (3)
Constitutional Symptoms (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Pulmonary/Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No